CLINICAL TRIAL: NCT07112872
Title: A Randomized, Double-Blind, Placebo- and Open-Label Active Comparator- Controlled, Parallel-Group, Multi-Center Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of Once-Daily RO7795081 Administered for 30 Weeks to Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Compare Different Doses of RO7795081 With a Placebo or Semaglutide in People With Type 2 Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP45703; 2024-520322-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Arm 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2: Semaglutide 14 mg (Active Comparator)
  Interventions: Drug: Semaglutide
- Arm 3: RO7795081 Dosing Regimen 1 (Experimental)
  Interventions: Drug: RO7795081
- Arm 4: RO7795081 Dosing Regimen 2 (Experimental)
  Interventions: Drug: RO7795081
- Arm 5: RO7795081 Dosing Regimen 3 (Experimental)
  Interventions: Drug: RO7795081
- Arm 6: RO7795081 Dosing Regimen 4 (Experimental)
  Interventions: Drug: RO7795081
- Arm 7: RO7795081 Dosing Regimen 5 (Experimental)
  Interventions: Drug: RO7795081
- Arm 8: RO7795081 Dosing Regimen 6 (Experimental)
  Interventions: Drug: RO7795081
- Arm 9: RO7795081 Dosing Regimen 7 (Experimental)
  Interventions: Drug: RO7795081

INTERVENTIONS:
Drug: RO7795081 — RO7795081 will be taken orally once daily (QD), according to the randomized dosing regimen, during the 30-week treatment period.
  Other Names: CT-996; RG6652
  Arms: Arm 3: RO7795081 Dosing Regimen 1; Arm 4: RO7795081 Dosing Regimen 2; Arm 5: RO7795081 Dosing Regimen 3; Arm 6: RO7795081 Dosing Regimen 4; Arm 7: RO7795081 Dosing Regimen 5; Arm 8: RO7795081 Dosing Regimen 6; Arm 9: RO7795081 Dosing Regimen 7
Drug: Semaglutide — Semaglutide 14 mg will be taken orally QD, with up-titration as per label, during the 30-week treatment period.
  Arms: Arm 2: Semaglutide 14 mg
Drug: Placebo — Placebo will be taken orally QD during the 30-week treatment period.
  Arms: Arm 1: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo- and open-label active comparator-controlled, parallel-group, dose-range-finding, Phase II study aims to evaluate the efficacy, tolerability, and safety of RO7795081 for glycemic control in adult participants with Type 2 diabetes mellitus (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type 2 diabetes mellitus (T2D) for at least 6 months before screening
* Have an HbA1c ≥7% and ≤10.5% at screening
* Management of T2D with diet and exercise alone or with either a stable dose of metformin or/and sodium-glucose cotransporter-2 (SGLT-2) inhibitors
* Body mass index (BMI) ≥23.0 kg/m^2 at screening
* A stable body weight within 3 months prior to screening (maximum 5% self-reported body weight gain and/or loss)

Exclusion Criteria:

* Have Type 1 diabetes (T1D), history of ketosis or hyperosmolar state/coma, or any other types of diabetes except T2D
* Have had 1 or more episodes of Level 3 hypoglycemia or has hypoglycemia unawareness within the 6 months prior to screening
* History or presence of proliferative diabetic retinopathy, diabetic macular edema, or non-proliferative diabetic retinopathy that requires acute treatment
* Evidence of clinically significant/active nephropathy or neuropathy (including resting tachycardia, orthostatic hypotension, and diabetic diarrhea)
* Current treatment or treatment within 3 months of screening with any other anti-hyperglycemic medication except metformin or SGLT-2 inhibitors
* Have obesity induced by other endocrinologic disorders (e.g., Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., melanocortin-4 receptor deficiency or Prader-Willi Syndrome)
* Have a known, clinically significant gastric emptying abnormality
* Have poorly controlled hypertension at screening, untreated renal artery stenosis, or evidence of labile blood pressure including symptomatic postural hypotension
* Have any of the following cardiovascular conditions within 3 months prior to screening: Acute myocardial infarction; Cerebrovascular accident (stroke)/transient ischemic attack; Unstable angina; Hospitalization due to congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-02-08 (Estimated); Study Completion 2027-02-08 (Estimated)

PRIMARY OUTCOMES:
RO7795081 vs. Placebo: Change in Glycated Hemoglobin (HbA1c) from Baseline at Week 30 | Baseline to Week 30

SECONDARY OUTCOMES:
RO7795081 vs. Semaglutide: Change in HbA1c from Baseline at Week 30 | Baseline to Week 30
Percentage of Participants with HbA1c <5.7%, ≤6.5%, and <7.0% at Week 30 | Week 30
Change in Fasting Plasma Glucose from Baseline at Week 30 | Baseline to Week 30
Percent Change in Body Weight from Baseline at Week 30 | Baseline to Week 30
Absolute Change in Body Weight (kg) from Baseline at Week 30 | Baseline to Week 30
Percentage of Participants Who Achieve ≥5%, ≥10%, or ≥15% Body Weight Reduction from Baseline at Week 30 | Baseline and Week 30
Incidence of Adverse Events (AEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) | From first dose until 28 days after the final dose of study treatment (34 weeks)
Number of Participants with Documented Hypoglycemia (Level 1, 2, or 3 per American Diabetes Association 2025) | From first dose until 28 days after the final dose of study treatment (34 weeks)
Plasma Concentrations of RO7795081 at Prespecified Timepoints | Predose on Day 1 and at prespecified timepoints until Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- United States (24):
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Orange County Research Center, Lake Forest, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research, Waterbury, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - K2 Medical Research South Orlando, LLC, Clermont, Florida
  - Center for Diabetes, Obesity and Metabolism Inc, Pembroke Pines, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Accellacare of Duly Health and Care, Oak Lawn, Illinois
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Accellacare of Piedmont Healthcare, Statesville, North Carolina
  - Accellacare of Wilmington, LLC, Wilmington, North Carolina
  - NexGen Research, Lima, Ohio
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Alliance for Multispecialty Research. LLC, Knoxville, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Apex Mobile Clinical Research, Bellaire, Texas
  - Velocity Clinical Research, Dallas, Texas
  - Velocity Clinical Research (Impact Research Institute), Waco, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
- Hungary (2):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Qualiclinic Kft., Budapest
- Poland (10):
  - NZOZ Osteo-Medic s.c. A. Racewicz, J.Supronik, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne INTERCOR Sp. z o.o., Bydgoszcz
  - Pro Familia Altera Sp z o.o., Katowice
  - ETG Lublin, Lublin
  - Ekamed sp. z o.o., Lublin
  - NZOZ METABOLICA O?rodek Bada? Klinicznych, Tarnów
  - ETG Warszawa, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
  - ETG Zamosc, Zamość
- Spain (15):
  - Universidad de Sevilla - Hospital Universitario Virgen Macarena, Seville, Barcelona
  - Instituto De Investigacion Marques De Valdecilla (IDIVAL), Santander, Cantabria
  - Hospital Vithas Nisa Sevilla, Castilleja de la Cuesta, Granada
  - Hospital Universitario A Coruna, A Coruña, LA Coruna
  - Complexo Hospitalario Universitario de Ferrol (CHUF), Ferrol, LA Coruna
  - Hospital Regional Universitario de Malaga, Malaga, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - centro Medico Teknon, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Hospital Clínico San Carlos, Madrid
  - Nuevas Tecnologias en Diabetes y Endocrinologia, Seville
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Clinico Universitario de Valencia (Instituto de Investigacion Sanitaria INCLIVA), Valencia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing